CLINICAL TRIAL: NCT02439944
Title: Efficacy and Neural Correlates of Personalized Treatment With Transdermal Nicotine Replacement: A Randomized, Controlled Pilot Study in Motivated Smokers Unable to Quit With Standard Dosing
Brief Title: Efficacy and Neural Correlates of Personalized Treatment With Transdermal Nicotine Replacement
Acronym: iT-NRT
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: full RCT funded. no need to continue pilot data collection.
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Laurie Zawertailo, Clinical Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 095/2014
Record Dates: First submitted 2015-05-07; First posted 2015-05-12 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Tobacco Use Disorder; Nicotine Dependence
Keywords: Nicotine Patch; Nicotine Mouth Spray; Smoking Cessation; Quit Smoking; Abstinence; Dependence; Nicotine; Tobacco; Transdermal Nicotine Replacement Therapy; Functional Magnetic Resonance Imaging; Neuroimaging; Cue Reactivity; Resting State; BOLD fMRI
MeSH Terms: conditions — Tobacco Use Disorder; Smoking Cessation | interventions — Tobacco Use Cessation Devices; Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Arm (Experimental): Escalating nicotine patch dose to satiety over 6 weeks with dosage depending on the number of cigarettes smoked per day and the occurrence of adverse effects
  Interventions: Drug: Nicotine patch
- Positive Control Arm (Active Comparator): Nicotine patch dose of 21mg coupled with nicotine mouthspray which is to be used as needed.
  Interventions: Drug: Nicotine patch; Drug: Nicotine mouthspray

INTERVENTIONS:
Drug: Nicotine patch
  Other Names: Nicoderm
Drug: Nicotine mouthspray
  Other Names: Nicorette Quickmist
  Arms: Positive Control Arm

SUMMARY:
This study involves the use of personalized nicotine patch dosing as a treatment strategy for smokers who cannot quit smoking after 2 weeks of using the standard nicotine patch dose. Functional Magnetic Resonance Imaging scans will also be obtained from all study participants before and after treatment. The first aim of the study is to determine if the treatment method under investigation is safe and more effective at increasing quit rates in smokers who do not respond to standard therapy.The second aim is to determine if there are any treatment- or cessation-related changes in brain function.

DETAILED DESCRIPTION:
Nicotine Replacement Therapy (NRT) is limited in efficacy. One possible explanation for this limited efficacy is that the nicotine dose received in standard therapy is not enough to replace the amount of nicotine that smokers typically receive from their cigarettes. In an effort to counteract this problem, this study will increase the nicotine patch dose of smokers until they no longer feel the need to keep smoking or they cannot tolerate a higher nicotine dose. Smokers who cannot quit using 21 mg nicotine patch for 2 weeks will be randomized to either the experimental arm of the study where nicotine patch doses will be adjusted according to individual need or the positive control arm where standard NRT smoking cessation therapy will be employed. The primary outcome measure will be continuous abstinence during the last 4 weeks of treatment. In addition, participants will be assessed to see how treatment has impacted their resting state neural activity as well as their responsiveness to smoking and emotional cues. Follow up sessions will be used to assess long term abstinence as well as long term change in neural activation.

ELIGIBILITY:
Inclusion Criteria:

* Daily tobacco smoker of
* Aged 19 to 65 years old
* Intending to quit smoking within the next 30 days
* Interested in using transdermal nicotine replacement therapy (nicotine patch)

Exclusion Criteria:

* At least weekly use of tobacco products other than cigarettes
* Breast feeding, pregnancy or not using a reliable form of birth control
* Any generalized skin disorders precluding the use of the patch
* Immediate post-myocardial infarction period or life-threatening arrhythmias, severe or worsening angina pectoris or recent cerebral vascular accident
* Any clinically significant electrocardiogram (ECG) abnormalities
* Currently using NRT or other smoking cessation pharmacotherapy
* Any known hypersensitivity or allergies to any of the components comprising the nicotine patch
* MRI contraindications (e.g., metal in body, claustrophobia) as per the CAMH RIC screening questionnaire
* Diagnosis of terminal illness.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
4 weeks continuous smoking abstinence | Treatment weeks 9-12 inclusive
  4 weeks of abstinence without a single puff of a cigarette confirmed by self-report and exhaled carbon monoxide (CO less than or equal to 4ppm)

SECONDARY OUTCOMES:
Cue induced brain activation | up to 6 month follow-up
  Brain activation in response to viewing emotional and smoking cues as measured by fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Zawertailo, PhD, Principal Investigator — Centre for Addiction and Mental Health; Peter Selby, MBBS, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Nicotine Dependence Clinic, Toronto, Ontario, Canada